CLINICAL TRIAL: NCT05199467
Title: A Pilot Trial of Health Coaching to Improve Functioning and Reduce Suicide Risk Among Reintegrating Veterans
Brief Title: Health Coaching: A Pilot Trial Among Reintegrating Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Michigan (Other); VA Finger Lakes Healthcare System (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: D3704-R
Record Dates: First submitted 2021-12-10; First posted 2022-01-20 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Veteran Reintegration
Keywords: Veterans; Vocational rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Health Coaching (Experimental): Receipt of up to 12 sessions of health coaching, plus printed materials providing information on VA benefits
  Interventions: Behavioral: Health Coaching; Behavioral: VA Benefits Information
- VA Benefits Information (Active Comparator): Receipt of printed materials providing information on VA benefits
  Interventions: Behavioral: VA Benefits Information

INTERVENTIONS:
Behavioral: Health Coaching — Health coaches help people focus on goals, identify strengths and values, and work towards building the kind of life they wish to live.
  Arms: Health Coaching
Behavioral: VA Benefits Information — Printed materials with information on VA benefits.

SUMMARY:
Health coaches help people focus on goals, identify strengths and values, and work towards building the life they wish to live. Health coaching may be especially helpful for people navigating a life transition, such as Veterans who recently separated from military service (i.e., reintegrating Veterans). In this pilot trial the investigators will 1) examine the feasibility of study procedures and acceptability of health coaching among reintegrating Veterans, 2) evaluate measures for suitability in a future trial that will examine efficacy of the intervention, 3) determine barriers and facilitators to implementing the intervention among reintegrating Veterans.

DETAILED DESCRIPTION:
This pilot study is designed to provide data to inform the design and procedures of a future efficacy trial of health coaching among reintegrating Veterans. An enrollment rate 30% and an assessment completion rate 65% at 9 months will be considered feasible enrollment and assessment completion rates for a future efficacy trial. An intervention completion rate 70% and mean score 27 on the Client Satisfaction Questionnaire-8 will indicate acceptability. Evaluation of measures will entail quantifying the mean levels in this population, characterizing typical variation in the outcomes, descriptive analyses of within-person change across time, and adjusted estimates of treatment effect sizes with 95% confidence intervals to calibrate the sample size needs of a fully powered trial. Qualitative interviews with participants will provide information on barriers and facilitators to implementation as well as perceived benefits and potential harms.

ELIGIBILITY:
Inclusion Criteria:

* United States military Veterans recently separated from service

Exclusion Criteria:

* Currently living in an institution (e.g., nursing home, prison)
* Cognitive impairment as indicated by a score equal to or greater than 10 on the Short Blessed Test
* Currently experiencing psychosis as indicated by endorsing thought interference or hallucinations on the Psychosis Screening Questionnaire
* At acute risk for suicide as indicated by the P4 screener
* Unable to read or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Military to Civilian Questionnaire | Month 4
  The Military to Civilian Questionnaire scores range from 0 to 4, with higher scores indicating a higher degree of reintegrating difficulty.
Well-being Inventory - Functional Status | Month 4
  The Functional Status composite measure from the Well-being Inventory scores range from 1 to 5, with higher scores indicating a higher level of functioning.
Military to Civilian Questionnaire | Month 9
  The Military to Civilian Questionnaire scores range from 0 to 4, with higher scores indicating a higher degree of reintegrating difficulty.
Well-being Inventory - Functional Status | Month 9
  The Functional Status composite measure from the Well-being Inventory scores range from 1 to 5, with higher scores indicating a higher level of functioning.
Depressive Symptom Index - Suicidality subscale | Month 4
  The Suicidality subscale of the Depressive Symptom Index scores range from 0 to 12, with higher scores indicating higher suicidal ideation severity.
Columbia Suicide Severity Rating Scale | Month 4
  The Columbia Suicide Severity Rating Scale - Screen scores range from 0 to 7, with higher scores indicating higher suicidal ideation severity.
Depressive Symptom Index - Suicidality subscale | Month 9
  The Suicidality subscale of the Depressive Symptom Index scores range from 0 to 12, with higher scores indicating higher suicidal ideation severity.
Columbia Suicide Severity Rating Scale | Month 9
  The Columbia Suicide Severity Rating Scale - Screen scores range from 0 to 7, with higher scores indicating higher suicidal ideation severity.

SECONDARY OUTCOMES:
Number of VA healthcare visits (primary care, mental health, or other specialty care visits) | Month 4
  Number of VA healthcare visits (primary care, mental health, or other specialty care visits) completed during the first four months of study participation, with higher number of visits indicating higher VA care utilization.
Number of VA healthcare visits (primary care, mental health, or other specialty care visits) | Month 9
  Number of VA healthcare visits (primary care, mental health, or other specialty care visits) completed during study participation (9 months), with higher number of visits indicating higher VA care utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M. Denneson, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT05199467/ICF_000.pdf